CLINICAL TRIAL: NCT02563886
Title: Electrically Assisted Movement Therapy (EAMT) for Upper Limb Stroke Rehabilitation
Brief Title: Electrically Assisted Movement Therapy
Acronym: EAMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Swiss Commission for Technology and Innovation (Other)
Responsible Party: Principal Investigator, Stefano Carda, MD, PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EAMT-346/15
Record Dates: First submitted 2015-09-22; First posted 2015-09-30 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EAMT, then standard care (Experimental): Electrically Assisted Movement Therapy precedes usual and customary care.
  Interventions: Other: Electrically Assisted Movement Therapy; Other: Usual and customary care
- Standard care, then EAMT (Active Comparator): Usual and customary care precedes Electrically Assisted Movement Therapy.
  Interventions: Other: Electrically Assisted Movement Therapy; Other: Usual and customary care

INTERVENTIONS:
Other: Electrically Assisted Movement Therapy — Electrically Assisted Movement Therapy (EAMT) is an extension of conventional Constraint-Induced Movement Therapy (CIMT) for moderately-to-severely paralyzed patients. During EAMT, patients use a movement controller with the healthy hand, controlling movements generated through neuromuscular electrical stimulation of the paralyzed arm and hand. During each session three types of exercises can be performed: mobilization, games, and training for activities of daily living, all three involving proper shaping of exercise difficulty at therapist discretion. Therapy consists in 20 sessions of 45 minutes twice per day over five weeks.
  Other Names: EAMT
Other: Usual and customary care — Usual and customary care ranges from no treatment to varying amounts of orthotics, home-based and clinic-based occupational therapy, or physiotherapy, but always excludes CIMT and EAMT. Therapy consists in 20 sessions of 45 minutes twice per day over five weeks, whenever possible, to match EAMT amount of therapy.
  Other Names: Standard care

SUMMARY:
The purpose of this study is to determine whether intensive, focused training of the affected upper extremity after stroke results in long-term functional gains in moderately-to-severely paralyzed patients, more than 6 months after their vascular accident. During the course of therapy, user's attempts to move and complete exercises are assisted by neuromuscular electrical stimulation.

DETAILED DESCRIPTION:
This pilot study quantifies functional gains induced by the Electrically Assisted Movement Therapy (EAMT), an extension of Constraint-Induced Movement Therapy to moderately-to-severely paralyzed patients in their stable plateau phase of recovery. During EAMT, patients can assist affected upper limb movements through functional electrical stimulation. Initially, patients are divided in two groups. One of the groups receives EAMT, the other receives the best possible physical and occupational therapy. Therapy consists in 40 sessions of 45 minutes twice per day over five weeks, including a one-week therapy break. After 20 sessions, group allocation is crossed-over, and patients don't receive any therapy for one week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one, first ever stroke (both ischemic or hemorrhagic) verified by brain imaging (MRI or CT);
* Chronic impairment after stroke (minimum 6 months);
* No contraindications to MRI;
* No contraindications to electrical stimulation;

Exclusion Criteria:

* Unstable recovery stage (difference between two examinations > 1 FMA-UE point);
* Mild impairment of the upper extremity (FMA-UE >= 21);
* Excessive spasticity of the affected arm (modified Ashworth Scale > 2);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment of the Upper Extremity (FMA-UE), | T0 (Before treatment); T1 (3 weeks after start and before treatment crossover); T2 (6 weeks after T0, at the end of treatment); T3 (3 months after treatment); T4 (6 months after treatment)
  A quantitative measure of motor impairment.

SECONDARY OUTCOMES:
Wolf Motor Function Test | T0 (Before treatment); T1 (3 weeks after start and before treatment crossover); T2 (6 weeks after T0, at the end of treatment); T3 (3 months after treatment); T4 (6 months after treatment)
  Quality and time of task performance
Modified Ashworth scale | T0 (Before treatment); T1 (3 weeks after start and before treatment crossover); T2 (6 weeks after T0, at the end of treatment); T3 (3 months after treatment); T4 (6 months after treatment)
  A quantitative measure of hand and arm spasticity
European stroke scale | T0 (Before treatment); T1 (3 weeks after start and before treatment crossover); T2 (6 weeks after T0, at the end of treatment); T3 (3 months after treatment); T4 (6 months after treatment)
  Overall functional status
Motor Activity Log | T0 (Before treatment); at 1, 2, 3, 4, 5, 6, 18 and 30 weeks after treatment start
  Semi-structured interview to assess arm function.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Carda, MD, PhD, Principal Investigator — Neuropsychology and Neurorehabilitation Service, Centre hospitalier universitaire vaudois (CHUV); José del R. Millán, Prof., Study Director — Defitech Foundation Chair in Brain-machine Interface, Swiss Federal Institute of Technology Lausanne (EPFL)
Locations (1):
- Service de Neuropsychologie et neuroréhabilitation - CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carda S, Biasiucci A, Maesani A, Ionta S, Moncharmont J, Clarke S, Murray MM, Millan JDR. Electrically Assisted Movement Therapy in Chronic Stroke Patients With Severe Upper Limb Paresis: A Pilot, Single-Blind, Randomized Crossover Study. Arch Phys Med Rehabil. 2017 Aug;98(8):1628-1635.e2. doi: 10.1016/j.apmr.2017.02.020. Epub 2017 May 9. PMID 28499657